CLINICAL TRIAL: NCT07076043
Title: Multi-product PrEP Delivery to Young Women Seeking Reproductive Health Services and Coverage of HIV Prevention
Acronym: PrEMIA
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: University of Washington (Other); Kenya Medical Research Institute (Other); National Institute of Mental Health (NIMH) (NIH); Partners in Health and Research Development (Unknown)
Responsible Party: Principal Investigator, Renee Heffron, Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: KEMRI/SERU/CCR/0361/5052; R01MH134681 (NIH)
Record Dates: First submitted 2025-07-17; First posted 2025-07-20 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: Hiv
Keywords: HIV prevention; PrEP; Adolescent girls and young women; Kenya; stepped wedge cluster randomized trial
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Standard of Care PrEP Program (No Intervention): In the control phase, clinics will offer standard of care PrEP program, which includes daily oral PrEP, for young women.
- Multiple Product PrEP Program (Active Comparator): In the intervention phase, clinics will offer a multi-product PrEP program, which includes daily oral PrEP and other forms of PrEP that are available. To start, the dapivirine vaginal ring will be included among the other forms of PrEP that are available. Others will be added as they become available in Kenya.
  Interventions: Drug: Multiple Product PrEP Program

INTERVENTIONS:
Drug: Multiple Product PrEP Program — In the intervention phase, clinics will offer a multi-product PrEP program, which includes daily oral PrEP and other forms of PrEP that are available. To start, the dapivirine vaginal ring will be included among the other forms of PrEP that are available. Others will be added as they become available in Kenya.
  Arms: Multiple Product PrEP Program

SUMMARY:
Following on the heels of large implementation science projects that participated in the launch of widespread daily oral PrEP availability, we will launch and study the integration of novel PrEP products - beginning with the dapivirine ring- into existing PrEP programs that reach women seeking reproductive health care at health facilities in Kenya. Intervention delivery will be launched among 12 participating clinics with approximately 1400 AGYW seeking reproductive health services and counseled about PrEP through a stepped wedge cluster randomized trial. We will support participating clinics to add dapivirine ring into their existing PrEP services offered to women seeking reproductive health care. Our primary aim will be to determine whether the availability of multiple PrEP products to young women will result in greater frequency of PrEP initiation and persistence.

ELIGIBILITY:
Inclusion Criteria for Adolescent Girls and Young Women seeking reproductive health services:

Age ≥18 years and ≤30years. Seeking a reproductive health service from one of the project facilities (reproductive health services include but are not limited to family planning, maternal and child health, postnatal care).

AGYW receiving reproductive health-related services through OPD, or other departments are eligible. AGYW receiving reproductive health-related services through other departments are eligible.

Willing and able to partake in an informed consent process. Able to speak and read in Kiswahili or English.

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Female
Enrollment: 1400 (Estimated)
Dates: Start 2025-06-03 (Actual); Primary Completion 2028-12-30 (Estimated); Study Completion 2029-12-30 (Estimated)

PRIMARY OUTCOMES:
PrEP initiation | From enrolment to 6 months
  Women who start to use PrEP

SECONDARY OUTCOMES:
PrEP persistence at 3 months | From enrolment to 3 months
  Women who continue to use PrEP 3 months since they initiated PrEP

OTHER OUTCOMES:
PrEP persistence at 6 months | Enrolment to 6 months
  Women who continue to use PrEP 6 months since they initiated PrEP

CONTACTS AND LOCATIONS:
Overall Officials: Nelly Mugo, MBChB, MMed, MPH, Principal Investigator — Kenya Medical Research Institute
Locations (1):
- Kenya Medical Research Institute and Partners in Health & Research Development, Thika, Kiambu County, Kenya

IPD SHARING:
Plan to Share IPD: Undecided